CLINICAL TRIAL: NCT05218967
Title: Virtual Reality as a Distraction Intervention for Pain Management During Office Laryngeal Procedures: Randomized Single Blinded Clinical Trial
Brief Title: Virtual Reality in Laryngology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-01021300
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pain Management During Office Laryngeal Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-office procedure with VR-assistance (Experimental)
  Interventions: Other: Virtual Reality Headset
- In-office procedure without VR-assistance (No Intervention)

INTERVENTIONS:
Other: Virtual Reality Headset — A head-worn apparatus that completely covers the eyes for an immersive 3D experience. The VR headset will be worn during the procedure.
  Arms: In-office procedure with VR-assistance

SUMMARY:
The purpose of this study is to compare patient's pain and anxiety undergoing laryngeal procedures and esophageal manometry while wearing a VR headset to standard of care. It is hypothesized that patient's using the VR headset during the procedure will have reduced pain and anxiety as compared to their standard of care counterparts because the VR environment will distract them from their procedure.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial, comparing patients' pain and anxiety experience while wearing a VR headset and receiving standard analgesia during In-office aerodigestive procedures (IOAEP) to patients' experience receiving standard analgesia only during IOAEP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 or older)
* Patients scheduled for IOAEP, including laryngeal biopsies, percutaneous injection laryngoplasty, KTP ablation of hemorrhagic polyps and respiratory papilloma, and transnasal esophagoscopy (TNE), and esophageal manometry.

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable to consent
* Non-English-speaking patients
* Patients who have undergone prior IOAEP
* Patients who have used any psychotropic or analgesic medication within the last 24 hours due to the possible confounding effect on pain or anxiety perception
* Patients with motion sickness or uncorrected visual impairment (legal blindness)
* Patients with past medical history of seizures or visual abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Pain during procedure, as measured by the McGill Pain Questionnaire | During Procedure
  individually rated pain descriptors with 11 addressing sensory pain and 4 focusing on affective components of pain. Each item is rated on a 4-point scale that ranges from none to severe.
Anxiety during the procedure , as measured by the spielberger State-Trait Anxiety Inventory (SF- STAI) | During Procedure
  The STAI consists of 6 questions concerning patient's current state of anxiety with responses ranging from (1) never to almost always (4).
Post Procedure Patient Questionnaire | Immediately After Procedure
  Patients will be asked if they would repeat the procedure again on a scale of 1-5 with 1 being never and 5 being always.
Physician Questionnaire | Immediately After Procedure
  Clinicians will fill out a short 6 question survey about the use of VR during their procedure. The survey is a short 6 item questionnaire inquiring about difficulty and success of the procedure, perceived patients' discomfort, observed patient agitation, interference and benefit of the VR headset. These questions will be answered using a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Heart rate | Measures will be recorded immediately before and immediately after the procedure.
  Heart rate will will be measured through AD instruments PowerLab.
Temperature | Measures will be recorded immediately before and immediately after the procedure.
  Temperature will be measured through AD instruments PowerLab
Galvanic Skin Activity | Measures will be recorded immediately before and immediately after the procedure.
  Galvanic Skin Activity will be measured through AD instruments PowerLab
Pain as measured by the Visual Analog Scale | Measures will be recorded immediately after the procedure.
  Visual Analog Pain Scale measured pain on range from 0-100 (0 is no pain and 100 is max pain) about time of pain, unpleasantness, average pain, and worst pain on a scale of 0-100.
Upper Esophageal Sphincter Pressure | During the Procedure
  Upper Esophageal Sphincter Pressure will be measured through the probe inserted during the High Resolution Manometry

CONTACTS AND LOCATIONS:
Overall Officials: Anais Rameau, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No